CLINICAL TRIAL: NCT04781114
Title: A Phase III, Randomized, Double-blind, Placebo-controlled Clinical Study Evaluating the Efficacy and Safety of JS002 in Patients With Primary Hypercholesterolemia and Mixed Hyperlipidemia in China
Brief Title: The Safety and Efficacy of Multiple-dose of JS002 in Subject With Hyperlipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JS002-003
Record Dates: First submitted 2021-02-24; First posted 2021-03-04 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2021-02

CONDITIONS: Hyperlipemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JS002 (Experimental): Cohort 1: 150 mg/1mL Q2W Subcutaneous(SC); Cohort 2: 300/2mL mg Q4W Subcutaneous(SC);
  Interventions: Drug: JS002
- Placebo (Placebo Comparator): Cohort 1: 1mL Q2W Subcutaneous(SC); Cohort 2: 2mL Q4W Subcutaneous(SC);
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JS002 — JS002: 150mg(1mL) Q2W; Placebo 1mL Q2W.
  Arms: JS002
Drug: Placebo — JS002: 300mg(2mL) Q4W; Placebo 2mL Q4W.
  Arms: Placebo

SUMMARY:
JS002 is a recombinant humanized anti-PCSK9 monoclonal antibody. This is a randomized, double-blind, placebo-controlled study to evaluate the safety and efficacy, as well as immunogenicity of JS002 treated repeatedly in patients with hyperlipidemia when combined with statin therapy.

In this study, two dose group (150 mg, 300 mg) were set up in this study. 750 subjects are plan to be enrolled (the study drug will be assigned to a 2:1 ratio of JS002 or placebo).

Each subject required a maximum of 6 weeks of screening, 52 weeks of treatment, and 8 weeks of follow-up.

ELIGIBILITY:
A limited list of criteria for selection of participants in the clinical study, provided in terms of inclusion and exclusion criteria and suitable for assisting potential participants in identifying clinical studies of interest. Use a bulleted list for each criterion below the headers "Inclusion Criteria" and "Exclusion Criteria". (Limit: 15,000 characters.) Inclusion criteria

1. Males and females ≥ 18 and ≤ 80 years of age;
2. LDL_C during screening period met the following conditions: super high risk: LDL - C ≥1.4mmol/L (55 mg/dL); extremely high risk: LDL - C ≥1.8 mmol/L (70 mg/dL); risk: LDL - C ≥2.6 mmol/L (100 mg/dL); low risk: LDL - C ≥ 3.4 /mmol/L (130 mg/dL)
3. Fasting triglycerides ≤4.5 mmol/L;

Exclusion criteria

1. Known HoFH;
2. History of NYHA class III-IV heart failure;
3. History of uncontrolled arrhythmia, Unstable angina,MI, PCI,CABG, DVT or pulmonary embolism within 3 months.
4. Uncontrolled hypertension.
5. Uncontrolled diabetes mellitius (HbA1c>8.0%）.
6. Other conditions that investigators considered inappropriate to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 806 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Change in LDL-C of JS002 | Up to 24Weeks after dose administration
  Percentage change in LDL-C relative to baseline at Week 24

SECONDARY OUTCOMES:
Change in LDL-C of JS002 | Up to 52Weeks after dose administration
  Percentage change in LDL-C relative to baseline at Week 52
Other lipid parameters of JS002 | Up to Week 24 and 52Weeks after dose administration
  Percentage change in LDL-C relative to baseline at Week 24 and Week 52
The occurrence of adverse events | Up 60Weeks after dose administration
  Evaluate the change of clinically significant laboratory tests, vital signs, and electrocardiogram
The immunogenicity of JS002 | Up 60Weeks after dose administration
  To evaluate the production time, duration and proportion of anti JS002 antibody (ADA).ADA positive samples are tested for titer and for neutralizing antibody (Nab).
Pharmacokinetics (PK) of JS002 | Up 60Weeks after dose administration
  Evaluation of Serum concentration of JS002.Descriptive statistics include mean (arithmetic mean and geometric mean), standard deviation (SD), coefficient of variation CV% (arithmetic coefficient and geometric coefficient of variation), Median (Median), minimum (Min) and maximum (Max).
Pharmacokinetics (PD) of JS002 | Up 60Weeks after dose administration
  Evaluation of serum concentrations of free/total PCSK9 and changes from baseline.Descriptive statistics include mean (arithmetic mean and geometric mean), standard deviation (SD), coefficient of variation CV% (arithmetic coefficient and geometric coefficient of variation), Median (Median), minimum (Min) and maximum (Max).

CONTACTS AND LOCATIONS:
Locations (57):
- China (57):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tongren Hospital Affiliated to Capital Medical University City:Beijing, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The 900 Hospital of the Joint Service Support Force of the People's Liberation Army of China, Fuzhou, Fujian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The First Hospital of Lanzhou University City:Lanzhou, Lanzhou, Gansu
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Guangdong General Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Hainan General Hospital, Haikou, Hainan
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Daqingshi People's Hospital, Daqing, Heilongjiang
  - The Fourth Affiliated Hospital of Harbin Medical University, Haerbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second People's Hospital of Changzhou, Changzhou, Jiangsu
  - Zhongda Hospital Southeast Universty, Nanjing, Jiangsu
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - The First Hospital of Nanchang, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - First Hospital of Jilin University, Changchun, Jilin
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - The central hospital of Dalian, Dalian, Liaoning
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - The People's Hospital of Liaoning Provincial, Shenyang, Liaoning
  - General Hospital of the PLA Northern Theater Command, Shenyang, Liaoning
  - Jinan Central Hospital, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - Xianyang Hospital of Yan 'an University, Xianyang, Shanxi
  - The First Affiliated Hospital of the Air Force Medical University, Xian, Shanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xian, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Teda International Cardiovascular Hospital, Tianjin, Tianjin Municipality
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang X, Qiu M, Cheng Z, Ji X, Chen J, Zhu H, Tang Y, Huang Z, Su G, Wang G, Huang Z, Yao Z, Lin J, Sun Y, Li S, Shao C, Zhao Y, Bai X, Han Y. Efficacy and Safety of Ongericimab in Chinese Patients With Primary Hypercholesterolemia and Mixed Dyslipidemia. J Am Heart Assoc. 2024 Jun 4;13(11):e033669. doi: 10.1161/JAHA.123.033669. Epub 2024 May 31. PMID 38818934